CLINICAL TRIAL: NCT03033641
Title: Feasibility of the CARTOFINDER™ 4D LAT Algorithm to Identify Ablation Target in Subjects With Atrial Fibrillation (FIND CAN Trial: "CF-172")
Brief Title: FIND CAN Trial: "CF-172"
Acronym: FIND CAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI CF-172
Record Dates: First submitted 2016-12-22; First posted 2017-01-27 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation procedure (Experimental)
  Interventions: Device: Ablation procedure

INTERVENTIONS:
Device: Ablation procedure — All enrolled subjects who have ablation targets identified will undergo CARTOFINDER guided ablation (CFGA) followed by PVI. Subjects will be followed per the protocol schedule. Subjects who have no ablation target identified on the baseline CARTOFINDER map will undergo ablation per the institution's standard of care and be followed for 7 days for safety monitoring, then exit from the study.
  Other Names: CARTOFINDER™ Workstation, CARTO® 3 EP Navigation System, with CARTOFINDER™ 4D LAT Algorithm installed (CARTOFINDER™ Module)

SUMMARY:
The purpose of this feasibility study is to further explore characteristics of ablation targets identified by CARTOFINDER 4D LAT Algorithm in subjects with persistent atrial fibrillation and to assess the acute outcome of CARTOFINDER Guided Ablation in terms of the termination of atrial fibrillation to either Normal Sinus Rhythm or Atrial Tachycardia.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following inclusion criteria:

1. Age > 18 years.
2. Patients who have signed the Patient Informed Consent Form (ICF)
3. Scheduled to undergo a clinically-indicated catheter ablation procedure for treatment of persistent atrial fibrillation (defined as continuous atrial fibrillation that is sustained beyond seven consecutive days).

   3.1. Drug-refractory atrial fibrillation. (failed 1 or more class I or III antiarrhythmic drugs) and demonstrating Persistent AF (requiring drugs or electrical shock to terminate)
4. Able and willing to comply with all pre-, post-, and follow-up testing and requirements (e.g. patients not confined by a court ruling)

Exclusion Criteria:

Subject who meet any of the following exclusion criteria are not eligible for enrollment.

1. Paroxysmal Atrial Fibrillation
2. Continuous AF > 12 months (1 Year) (Longstanding Persistent AF) 2.1. Subjects previously diagnosed as Long Standing Persistent (LSP) but have demonstrated the ability to maintain Normal Sinus Rhythm for >30 days after cardioversion and have not been in AF greater than 1 year at the time of the procedure remain eligible for inclusion.
3. Previous ablation procedure for AF (previous ablation for the treatment of Flutter is acceptable)
4. Patients with a left atrial size >55 mm (echocardiography, parasternal long axis view).
5. Inability to restore sinus rhythm for 30 seconds or longer in the opinion of the investigator.
6. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
7. Atrial arrhythmia patients with structural atrial disease such as a prior history of atriotomy from prior atrial surgery, presence of an atrial septal defect, and/or presence of an atrial septal closure patch.
8. History of or current blood clotting or bleeding abnormalities, contraindication to systemic anticoagulation (i.e., heparin, warfarin, dabigatran, or a direct thrombin inhibitor), significant pulmonary disease, unstable angina, uncontrolled heart failure, acute illness or systemic infection, or any other disease or malfunction that would preclude treatment in the opinion of the investigator.
9. Enrollment in a study evaluating another device or drug.
10. A complex arrhythmia secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
11. Patients with a prosthetic mitral valve or any mechanical valve
12. Any cardiac surgery within the past 60 days (2 months) (includes PCI) (bypass within the past year)
13. Subjects that have ever undergone valvular cardiac surgical procedure (ie, ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve)
14. Prior ICD or pacemaker implanted
15. Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction or manipulation.
16. Presence of a condition that precludes vascular access.
17. Subject has a contra-indication to any of the devices used in the study per the IFU
18. Women of child bearing potential who are pregnant, lactating, or planning to become pregnant during the course of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Evaluate mapping characteristics | Intraoperative
  Explore characteristics of ablation targets identified by the CARTOFINDER 4D LAT Algorithm
Evaluate acute safety of freedom from procedure-related primary adverse events | Within 7 days
  Evaluate acute safety of freedom from procedure-related primary adverse events occurring within 7 days of ablation procedure

SECONDARY OUTCOMES:
Evaluate atrial fibrillation (AF) termination | Perioperative
  Evaluate the AF termination to Normal Sinus Rhythm (NSR) or an Atrial Tachycardia (AT) after CARTOFINDER™ Guided Ablation (CFGA) of identified ablation target and after PVI

IPD SHARING:
Plan to Share IPD: No